CLINICAL TRIAL: NCT05580133
Title: All-Inside Single-Bundle for ACL Reconstruction With Full Thickness of the Peroneus Longus Tendon Compared to the Six-strand-hamstring Autograft
Brief Title: All-Inside Single-Bundle for Anterior Cruciate Ligament Reconstruction With Full Thickness of the Peroneus Longus Tendon Compared to the Six-strand-hamstring Autograft (ACL)
Acronym: ACL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, mohamed hedi ezzine, Principal Investigator, medical doctor, assistant professor, Mongi Slim Hospital
Other Study IDs: mongislim
Record Dates: First submitted 2022-09-27; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; peroneus longus tendon; Hamstring Tendons; donor site
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peroneus Longus Tendon autograft: All-Inside Single-Bundle for ACL Reconstruction with Full Thickness of the Peroneus Longus Tendon
  Interventions: Procedure: anterior cruciate ligament reconstruction
- six-strand-hamstring autograft: All-Inside Single-Bundle for ACL Reconstruction with six-strand-hamstring autograft
  Interventions: Procedure: anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: anterior cruciate ligament reconstruction — Arthroscopic reconstruction of the anterior cruciate ligament is a surgical tissue graft replacement of the anterior cruciate ligament, located in the knee, to restore function after injury.

SUMMARY:
Anterior cruciate ligament reconstruction is the current gold standard for restoring knee stability. Hamstring tendon (HT) autograft is the most popular graft choice for ACL reconstruction worldwide. Other autografts include bone-patellar tendon-bone and quadriceps tendon, yet no globally accepted gold standard of graft choice exists for use in ACL reconstruction.

The peroneus longus tendon (PLT) has been reported as an autograft choice for ligament reconstruction[2], but there is little information regarding the clinical outcomes using the peroneus longus tendon (AHPLT) compared with hamstring tendon autograft. Therefore, we are interested in investigating whether the clinical outcomes of the PLT autograft were equivalent to the Six-strand- hamstring tendon autograft.

DETAILED DESCRIPTION:
prospective randomized clinical study to compare the results of all-inside anatomical ACL reconstruction using the AHPLT and using Six-strand- tendon autograft.

Randomization will be done with inclusion criteria of primary ACL rupture in adult patients and exclusion criteria of serious osteoarthritis, revision cases, and multiple ligament injuries.

Preoperatively, physical examinations including the anterior drawer test and the pivot shift Test were performed to judge the stability of the knee joint. All of the patients will be evaluated with an International Knee Documentation Committee (IKDC) 2000 subjective score, a Visual Analogue Scale (VAS), and an American Orthopedic Foot and Ankle Score (AOFAS).a knee joint arthrometers was also used with knee flexion of 30° at 134 N.

All of the tests will be performed three times by another experienced orthopedic surgeon who is not involved in the surgery, and the mean of the three measurements will be taken as the final value.

ELIGIBILITY:
Inclusion Criteria:

* primary ACL rupture in adult patients

Exclusion Criteria:

* serious osteoarthritis
* revision cases
* multiple ligament injuries
* ankle injuries

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: study population is a young athletic population with anterior laxity of the knee secondary to anterior cruciate ligament injury
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
the anterior drawer test | Baseline,
  the anterior drawer test is used to assess the integrity of the anterior cruciate ligament. With the knee flexed to 90 degrees, the foot is stabilized by sitting on it. The proximal tibia is grasped firmly with both hands, and the tibia is forcibly pulled anteriorly, noting any or abnormal movement compared with the opposite side.
  to estimate how severe the injury is by how far they can displace the ACL. They grade the tear from one to three (I, II, or III), with three being the worst tear. A grade I tear moves 5 millimeters, a grade II tear moves between 5 and 10 millimeters, and a grade III tear moves more than 10 millimeters.
the anterior drawer test | Month 8
  the anterior drawer test is used to assess the integrity of the anterior cruciate ligament. With the knee flexed to 90 degrees, the foot is stabilized by sitting on it. The proximal tibia is grasped firmly with both hands, and the tibia is forcibly pulled anteriorly, noting any or abnormal movement compared with the opposite side.
  to estimate how severe the injury is by how far they can displace the ACL. They grade the tear from one to three (I, II, or III), with three being the worst tear. A grade I tear moves 5 millimeters, a grade II tear moves between 5 and 10 millimeters, and a grade III tear moves more than 10 millimeters.
The pivot shift | Baseline
  The pivot shift is a dynamic but passive test of knee stability, carried out by the examiner without any activity of the patient. It shows a dysregulation between rolling and gliding in the knee joint. The patient lies in supine. The movement is a combination of axial load and valgus force, applied by the examiner, during a knee flexion from an extended position. When the test is positive, it indicates an injury of the anterior cruciate ligament
The pivot shift | Month 8
  The pivot shift is a dynamic but passive test of knee stability, carried out by the examiner without any activity of the patient. It shows a dysregulation between rolling and gliding in the knee joint. The patient lies in supine. The movement is a combination of axial load and valgus force, applied by the examiner, during a knee flexion from an extended position. When the test is positive, it indicates an injury of the anterior cruciate ligament
Visual Analogue Scale (VAS) | Baseline
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Visual Analogue Scale (VAS) | Week 3
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
International Knee Documentation Committee (IKDC) 2000 subjective score | Baseline
  The score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
International Knee Documentation Committee (IKDC) 2000 subjective score | Month 8
  The score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
knee joint arthrometers | Baseline
  a value less than 3 mm means that there is no ACL injury difference residing between 3 and 5 mm, it is considered that anterior posterior laxity is unusually high. The ACL might therefore be partially or completely torn.
  difference higher than 5 mm, it is considered that anterior posterior laxity is very high which indicates a complete ACL tear.
knee joint arthrometers | Month 8
  a value less than 3 mm means that there is no ACL injury difference residing between 3 and 5 mm, it is considered that anterior posterior laxity is unusually high. The ACL might therefore be partially or completely torn.
  difference higher than 5 mm, it is considered that anterior posterior laxity is very high which indicates a complete ACL tear.